CLINICAL TRIAL: NCT00391131
Title: A Multi-centre, Open-label Study to Assess the Efficacy, Tolerability, Safety and Pharmacokinetics of Subcutaneous Infusions of Ig NextGen 16% in Patients With Primary Immunodeficiency (PID).
Brief Title: Subcutaneous Ig NextGen 16% in PID Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CSL Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSLCT-SCIG-05-23
Record Dates: First submitted 2006-10-20; First posted 2006-10-23 (Estimated); Last update posted 2012-06-07 (Estimated); Status verified 2012-06

CONDITIONS: Primary Immunodeficiency (PID)
Keywords: PID; SCIG; Ig; Quality of Life; Serious Bacterial Infections
MeSH Terms: conditions — Primary Immunodeficiency Diseases

ARMS (1):
- Ig NextGen 16% (Experimental)
  Interventions: Drug: IgNextGen 16%

INTERVENTIONS:
Drug: IgNextGen 16% — IgNextGen 16% administered subcutaneously on a weekly basis from visit 1 to 12

SUMMARY:
This study aims to assess the safety, tolerability, efficacy and pharmacokinetics of Ig NextGen 16% in people with antibody deficiency currently being treated with IntragamP. Ig NextGen 16% is a liquid immunoglobulin (antibody) preparation manufactured using predominately chromatographic techniques. Eligible patients will switch from monthly intravenous IntragamP therapy to weekly subcutaneous Ig NextGen 16% treatment. Initial hospital training will be required for subcutaneous administration and then the patient will perform the infusion in their own home, returning once a month for a supervised infusion. Patients will be monitored on the study for up to 10 months to assess blood IgG levels and rate of serious bacterial infections.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:

  * Males or females 3 years of age or greater and at least 13 kg at enrolment.
  * PID patients receiving Ig replacement therapy, with a diagnosis of X-linked agammaglobulinemia (XLA) or Common Variable immunodeficiency (CVID) with severe hypogammaglobulinemia.
  * Patients who have received a consistent dose of Intragam®P at 3-, 4-, 5- or 6-weekly intervals, within the range of 0.2 - 0.6 g/kg body weight, for at least six months prior to the Screening visit.
  * Patients must have maintained IgG trough serum level of ≥ 5 g/L during the six months prior to Visit 0, with at least two trough levels to have been documented during this period.
  * Patients and/or their legally acceptable representative/guardian must give written informed consent to participate in the study and must understand the nature of the study and must be willing to comply with all protocol requirements

Exclusion Criteria:

* • Patients newly diagnosed with PID within six months of the Screening visit.

  * Patients with known or suspected severe hypersensitivity or previous evidence of severe side effects to immunoglobulin therapy or other blood products
  * Patients with known selective IgA deficiency or antibodies to IgA
  * Patients receiving immunosuppressive treatment other than topical and/or inhaled steroids and low dose oral steroids.
  * Females who are pregnant, breast feeding or planning a pregnancy during the course of the study. Females who are of child bearing potential must have a negative pregnancy test at screening.
  * Patients with protein-losing enteropathies, and kidney diseases with substantial proteinuria
  * Patients with malignancies of lymphoid cells such as chronic lymphocytic leukaemia, Non-Hodgkin's lymphoma and immunodeficiency with thymoma.
  * Patients who have within 30 days priors to the study screening visit, participated in a clinical study or used an investigational compound (eg: a new chemical entity not registered for clinical use).
  * Patients with any of the following abnormal lab results:

    * Serum creatinine >1.5 x Upper limit of Normal (ULN).
    * Serum ALT & AST > 2.5 x ULN.
    * Albumin < 25 g/L
  * Patients who are suffering from an acute or chronic medical condition, other than PID, which may, in the opinion of the Investigator, affect the conduct of the trial.
  * Patients who are not willing or are unable to comply with protocol.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2007-04; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Efficacy | Continually from Visits 7 to 12 & monthly IgG troughs

SECONDARY OUTCOMES:
Safety, Tolerability, Quality of Life, Pharmacokinetics | Visits 0, 6, 9, and12

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Empson, Dr, Principal Investigator — Auckland City Hospital
Locations (12):
- Australia (8):
  - The Canberra Hospital, Garran, Australian Capital Territory
  - John Hunter Hospital, New Lambton Heights, New South Wales
  - Sydney Children's Hospital, Randwick, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Women's & Children's Hospital, North Adelaide, South Australia
  - Frankston Hospital, Frankston, Victoria
  - Royal Children's Hospital, Melbourne, Victoria
  - Princess Margaret Hospital for Children, Perth, Western Australia
- New Zealand (4):
  - Auckland Hospital, Auckland
  - Starship Children's Hospital, Auckland
  - Christchurch Hospital, Christchurch
  - Wellington Hospital, Wellington

REFERENCES:
- [Result] Empson MB, Tang ML, Pearce LK, Rozen L, Gold MS, Katelaris CH, Langton D, Smart J, Smith WB, Steele RH, Ziegler JB, Maher D. Efficacy, safety and pharmacokinetics of a novel subcutaneous immunoglobulin, Evogam(R), in primary immunodeficiency. J Clin Immunol. 2012 Oct;32(5):897-906. doi: 10.1007/s10875-011-9641-4. Epub 2012 Apr 13. PMID 22526590